CLINICAL TRIAL: NCT01093157
Title: A Dose-finding Pilot Study of ACTH (Adrenocorticotropic Hormone) on the Proteinuria and Serum Lipoprotein Profile in Patients With Idiopathic Membranous Nephropathy (MN)
Brief Title: A Dose Escalation Study of Long-acting ACTH Gel in Membranous Nephropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-006328-GN; Health Canada (Registry Identifier: Health Canada 4727-88\3-23 C., control 131403)
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2013-01

CONDITIONS: Glomerulonephritis
Keywords: Kidney disease, Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis; Kidney Diseases | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACTH (HP Acthar gel) 40 units (Active Comparator)
  Interventions: Drug: Adrenocorticotrophic hormone ACTH
- ACTH (HP Acthar gel) 80 units (Active Comparator)
  Interventions: Drug: Adrenocorticotrophic hormone ACTH

INTERVENTIONS:
Drug: Adrenocorticotrophic hormone ACTH — There will be two arms to the study: one arm receive 40 units and the second arm 80 units of the ACTH gel subcutaneously both given in a dose escalating frequency beginning at once every two weeks escalating to a maximum of twice per week over a total of three months exposed.An ammendment(approved by Health Canada and the UHN IRB allows an additional 1 month of the perscribed therapy of ACTH )if there is an improvement in proteinuria at the end of the 3 month exposure.
  Other Names: HP Acthar gel

SUMMARY:
Membranous Nephropathy (MN) is an immune-mediated kidney disease that affects the glomerulus or the filter that removes toxins from the blood. Damage to the membrane that separates blood from urine results in loss of protein into the urine (proteinuria) and in some cases loss of kidney function.There is no standard specific treatment for MN.

ACTH has a pronounced lipid-lowering effect in healthy individuals, in steroid-treated patients with renal disease and in hemodialysis patients Some studies suggest that prolonged synthetic ACTH therapy may represent an effective therapy in patients with idiopathic MN, more extensive randomized studies with longer follow-up are needed before therapeutic recommendations can be made.

We propose to do a pilot study to test the hypothesis that biologic ACTH, a slow-release formulation of corticotropin extracted from porcine pituitary glands (H.P. Acthar gel) will be effective in reducing proteinuria and improving lipid profile in patients with idiopathic MN.

ELIGIBILITY:
Inclusion Criteria:• Idiopathic MN with diagnostic biopsy performed less than 36 months from the time of dose randomization.

* Patients need to be treated with an ACEI and/or ARB, for at least 3 months prior to ACTH treatment and have adequately controlled blood pressure (BP <130/75 mm Hg in >75% of the readings). Patients with documented evidence of >3 months treatment with maximal Ang II blockade, target BP (BP <130/75 mm Hg in >75% of the readings) and who remain with proteinuria >4.0g/24h may enter the ACTH phase of the study without the need to have the run-in/conservative phase of the study.
* Proteinuria as measured by Uprot/Ucr > 4.0 on a spot sample aliquot from a 24-hour urine collection. The choice of Uprot/UCr is in accord with recent NKF-CKD guidelines.[9]
* Estimated GFR ≥ 40 ml/min/1.73m2 while taking ACEI/ARB therapy. The GFR will be estimated using the 4 variable MDRD equation as published in the NKF-CKD guidelines.[9] The same NKF-CKD guidelines also promote the use of estimated GFR (GFRest) values rather than serum creatinine levels or CrCl measurements as the preferred non-invasive method of determining glomerular filtration rates.[9]

Exclusion Criteria:• Age <18 years.

* Estimated GFR < 40 ml/min/1.73m2, or serum creatinine >2.0 mg/dl.
* Renal biopsy showing more than 30% glomerulosclerosis and/or tubular atrophy.
* Patient must be off glucocorticoid, calcineurin inhibitors (cyclosporin A, tacrolimus) or mycophenolic mofetil for > 1 month, and alkylating agents or rituximab for >6 months.
* Resistance to the following immunosuppressive routines e.g. steroids alone, calcineurin inhibitors plus or minus steroids, cytotoxic agents plus or minus steroids.
* Patients with active infections or secondary causes of MN (e.g. hepatitis B, SLE, medications, malignancies). Testing for HIV, Hepatitis B and C should have occurred < 2 years prior to enrollment into the study.
* Type 1 or 2 diabetes mellitus: to exclude proteinuria secondary to diabetic nephropathy. Patients who have recent history of steroid induced diabetes but no evidence on renal biopsy performed within 6 months of entry into the study are eligible for enrollment.
* Pregnancy or nursing - for safety reasons.
* Acute renal vein thrombosis documented prior to entry by renal US or CT scan and requiring anticoagulation therapy.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-02; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
change in proteinuria from baseline to value at 3 months . | 3 months

SECONDARY OUTCOMES:
Complete Remission(CR) or Partial Remission (PR) at 3 months | 3 months
  Definition of proteinuric status. UP = urinary protein (g/24h) Complete remission (CR) UP ≤ 0.3 g Partial remission (PR) Reduction in UP of > 50% plus final UP ≤ 3.5 g but >0.3g Non-response (NR) Reduction in UP of < 50%. (includes increase in UP <50%) Progression Proteinuria increases by > 50%
Adverse effects | Throughout three months of this study and for nine months follow-up
  Patients will be directly questioned every two weeks during the drug exposure and then at monthly intervals during follow-up. In addition a contact number will be provided to the subjects to call if they experience any adverse affect or if they suspect adverse effect at any time between specific visits

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cattran, M.D, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952